CLINICAL TRIAL: NCT03645317
Title: A Study Investigating How to Avoid Cardiac Toxicity in Lung Cancer Patients Treated With Curative-intent Radiotherapy to Improve Survival, Funded by Yorkshire Cancer Research
Brief Title: Avoiding Cardiac Toxicity in Lung Cancer Patients Treated With Curative-intent Radiotherapy
Acronym: ACCOLADE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Prof Corinne Faivre-Finn (Other)
Collaborators: The Leeds Teaching Hospitals NHS Trust (Other); University of Manchester (Other); University of Leeds (Other); Manchester University NHS Foundation Trust (Other Government)
Responsible Party: Sponsor-Investigator, Prof Corinne Faivre-Finn, Professor of thoracic radiation oncology, The Christie NHS Foundation Trust
Organization: The Christie NHS Foundation Trust (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: M401
Record Dates: First submitted 2018-07-20; First posted 2018-08-24 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2021-07

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Hematologic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Other): Blood samples (FBC, lipids, cholesterol, troponin, CRP, BNP) Cardiac imaging (cardiac CT, cardiac ultrasound, 12-lead ECG)
  Interventions: Diagnostic Test: Blood tests & cardiac imaging

INTERVENTIONS:
Diagnostic Test: Blood tests & cardiac imaging — Blood tests (full blood count, lipids, cholesterol, high sensitivity Troponin levels, C-reactive protein (CRP) and brain natriuretic peptide) Cardiac imaging - cardiac CT, cardiac ultrasound, 12-lead ECG

SUMMARY:
Radiotherapy plays a major role in the treatment of lung cancer and recent advances in radiotherapy have led to better cure rates. However, the radiotherapy dose needed to destroy the cancer cells can unfortunately also damage the surrounding organs, such as the heart. The precise mechanism of damage and which areas of the heart are more sensitive to radiation is not currently known. This project uses the analysis of large amounts of existing radiotherapy treatment data to determine this. Establishing detailed radiotherapy dose limits for the heart and the heart's sub-structures will lead to the delivery of heart-sparing radiotherapy, where possible, in lung cancer patients treated in Yorkshire and Greater Manchester. The investigators estimate that this should lead to an improvement in one-year survival of approximately 10%.

ELIGIBILITY:
Inclusion Criteria:

* Histological or clinical diagnosis of lung cancer (Stage I-III non-small cell and small cell lung cancer) suitable for curative-intent radiotherapy
* Patients suitable for curative-intent radiotherapy (minimum 20 fractions for conventional fractionation and 3-8 fractions for SABR)
* Life expectancy > 4 months
* Age ≥ 18 years
* Patient has read and understood the participant information sheet and given informed consent

Exclusion criteria:

* No histological or clinical diagnosis of lung cancer (Stage I-III non-small cell and small cell lung cancer) and not suitable for curative-intent radiotherapy
* Patients not suitable for curative-intent radiotherapy (minimum 20 fractions for conventional fractionation and 3-8 fractions for SABR)
* Life expectancy < 4 months
* Age < 18 years
* Patient has not read and understood the participant information sheet and has not given informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-06-12 (Actual); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
The effect of radiation dose to the heart assessed using blood test (full blood count) | 4 months (duration of each participant on study)
  The effect of radiation dose to the heart assessed using full blood count measurement at the following time points (before radiotherapy, within 7 days post-radiotherapy and at 4 months post-radiotherapy)
The effect of radiation dose to the heart assessed using blood test (lipids & cholesterol - LDL & HDL levels) | 4 months (duration of each participant on study)
  The effect of radiation dose to the heart assessed using lipid & cholesterol (LDL & HDL) measurements at the following time points (before radiotherapy, within 7 days post-radiotherapy and at 4 months post-radiotherapy)
The effect of radiation dose to the heart assessed using blood test (troponin) | 4 months (duration of each participant on study)
  The effect of radiation dose to the heart assessed using troponin measurement at the following time points (before radiotherapy, within 7 days post-radiotherapy and at 4 months post-radiotherapy)
The effect of radiation dose to the heart assessed using blood test (C-reactive protein) | 4 months (duration of each participant on study)
  The effect of radiation dose to the heart assessed using C-reactive protein measurement at the following time points (before radiotherapy, within 7 days post-radiotherapy and at 4 months post-radiotherapy)
The effect of radiation dose to the heart assessed using blood test (brain natriuretic peptide) | 4 months (duration of each participant on study)
  The effect of radiation dose to the heart assessed using brain natriuretic peptide measurement at the following time points (before radiotherapy, within 7 days post-radiotherapy and at 4 months post-radiotherapy)
The effect of radiation dose to the heart assessed using cardiac imaging (cardiac ultrasound) | 4 months (duration of each participant on study)
  The effect of radiation dose to the heart assessed using cardiac ultrasound scans at the following time points (before radiotherapy and at 4 months after radiotherapy). The following components of the cardiac ultrasound measured during the study: parasternal long axis, parasternal short axis, apical 2/4/5 chambers, apical long axis, subcostal and parasternal notch.
The effect of radiation dose to the heart assessed using cardiac imaging (cardiac CT) | 4 months (duration of each participant on study)
  The effect of radiation dose to the heart assessed using cardiac CT scans at the following time points (before radiotherapy and at 4 months after radiotherapy). The following components of the cardiac CT scan measured during the study: coronary calcium score (Agaston/Volume) - CAC-RDS 0, CAC-RDS 1, CAC-RDS 2, CAC-RDS 3, CAC-RADS classification.
The effect of radiation dose to the heart assessed using cardiac imaging (12-lead ECG) | 4 months (duration of each participant on study)
  The effect of radiation dose to the heart assessed using 12-lead ECG at the following time points (before radiotherapy and at 4 months after radiotherapy). The following components of the ECG measured during the study: heart rate, rhythm, P wave, QRS complex, QT interval, ST segment & PR interval.

CONTACTS AND LOCATIONS:
Overall Officials: Corinne Faivre-Finn, PhD, Principal Investigator — The Christie NHS Foundation Trust / Univerrsity of Manchester
Locations (2):
- United Kingdom (2):
  - Leeds Teaching Hospitals NHS Trust, Leeds
  - The Christie NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: No
No plans to share data